CLINICAL TRIAL: NCT03051841
Title: A Phase I, Open-Label, Multi-Center Study of CKD-581 in Combination With Bortezomib and Dexamethasone in Patients With Previously Treated Multiple Myeloma
Brief Title: CKD-581 + Bortezomib + Dexamethasone in Patients With Previously Treated Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 133MM16010
Record Dates: First submitted 2017-01-09; First posted 2017-02-14 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Myeloma, Multiple
MeSH Terms: conditions — Multiple Myeloma | interventions — CKD-581

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treat Regimen (Experimental): CKD-581(investigational Drug) Bortezomib Dexamethasone
  Interventions: Drug: CKD-581

INTERVENTIONS:
Drug: CKD-581 — Intravenously on Days 1, 8 of each 21-day treatment cycle.
  Other Names: CKD-581 bortezomib dexamethasone regimen

SUMMARY:
This study is to determine the maximum tolerated dose(MTD), dose limiting toxicity(DLT), safety and pharmacokinetics(PK) profile of a single agent CKD-581 injection in Combination with Bortezomib and Dexamethasone in patients with Previously Treated Multiple Myeloma.

DETAILED DESCRIPTION:
This is an open label, dose escalation study. Cohort of 3~6 patients receive escalation doses of CKD-581 until the maximum toleated dose(MTD) is determined. The MTD is defiend as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* must have received at least one prior lines of therapy and Diagnosis of symptomatic multiple myeloma(IMWG 2014)
* Eastern Cooperative Oncology Group performance status ≤ 2
* Life expectancy 12 weeks
* must have the following laboratory values within 3 weeks prior to first dose of study drug

  * ANC(absolute neutrophil count) ≥ 1,500 mm3
  * PLT(platelet count)≥ 100,000 mm3
  * Hb ≥ 8.0g/dL
  * AST(SGOT) and ALT (SGPT) ≤ 3 x UNL(upper limit of normal)
  * Serum bilirubin ≤ 1.5 x ULN (but, Gilbert syndrome ≤ 3 x UNL)
  * Serum Cr ≤ 1.5 x UNL
* One more measureable disease following values

  * Serum M-protein ≥ 1g/dL
  * Urine M-Protein ≥ 200mg/24hr
  * in that case serum M-protein, urine M-Protein nonmeasurable and FLC ratio abnormal, Serum FLC level ≥ 100mg/L(≥10mg/dL)
* more than 24 weeks prior to last bortezomib dose
* must have signed the consent form

Exclusion Criteria:

* Patients with central neurological disease
* Patients with clinically significant heart disease within 24weeks prior to first dose of study drug
* patients with clinically significans abnormal EKG, echocardiography at screening
* patients with active hepatitis, HIV positive(exception, non active hepatitis)
* peripheral neuropathy ≥ CTCAE grade 2 or peripheral neuropathy ≥ CTCAE grade 1 with pain within 2 weeks prior to first dose of study drug
* Patients with a prior malignancy with in the last 3 years except adequately treated basal cell or squamous cell or skin cancer, in situ cervical cancer
* Patients who have received surgery, chemotherapy, radiation therapy or immunotherapy or any other investigational drugs ≤ 4 weeks prior to first dose of study drug and during treatment period
* Women who are pregnant or breast feeding or women of childbearing potential not using an effective method of birth control. Male patients whose sexual partners are not using effective birth control.
* patients with hypersensitive reaction of bortezomib or dexamethasone
* patients without best overall response is above minimal response based on IMWG 2015 past all treatment for multiple myeloma
* patients with refractory to past bortezomib treatment(ex; under minimal response) or progress within 60days prior to last bortezomib treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-04 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) | Up to 21 days(for 1st cycle)

SECONDARY OUTCOMES:
Pharmacokinetics(Cmax) | 1st Cycle day1, Day8: up to 24hr
Number of participants with toxicity as assessed by CTCAE v4.03 through study completion, an average of 1 year | through study completion, an average of 1 year
Objective Response Rate(ORR) of participants as assessed by IMWG uniform response criteria(2011) every 6weeks | every 6weeks, up to 1year
Progression Free Survival(PFS) of participants as assessed by IMWG uniform response criteria(2011) every 6weeks | Average time period between the start day of induction therapy and the day of relapse or progression or death, whichever occurs firstly, up to 1year
Overall Survival(OS) of participants as assessed by IMWG uniform response criteria(2011) every 6weeks | Average time period between the start day of induction therapy and the day of death, due to any cause, up to 1year
Duration of Response(DOR) of participants as assessed by IMWG uniform response criteria(2011) every 6weeks | Average time period between the day of first achievement of response and the day of first relapse or progression, up to 1year
Pharmacokinetics(T1/2) | 1st Cycle day1, Day8: up to 24hr
Pharmacokinetics(CL) | 1st Cycle day1, Day8: up to 24hr
Pharmacokinetics(AUClast) | 1st Cycle day1, Day8: up to 24hr
Pharmacokinetics(AUCinf) | 1st Cycle day1, Day8: up to 24hr
Pharmacokinetics(Vd) | 1st Cycle day1, Day8: up to 24hr
Pharmacokinetics( MRT) | 1st Cycle day1, Day8: up to 24hr

CONTACTS AND LOCATIONS:
Overall Officials: Min Ji Song, Study Director — Chong Kun Dang Pharmaceutical Corp.
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided